CLINICAL TRIAL: NCT06870565
Title: A Multicenter Randomized Study Comparing Paclitaxel and Platinum-based Concurrent Chemoradiotherapy With Short-term Adjuvant Chemotherapy Versus Platinum-based Monotherapy Concurrent Chemoradiotherapy in Patients With Postoperative Cervical Gastric-type Adenocarcinoma With High-risk Factors for Recurrence.
Brief Title: Comparative Study of Adjuvant Therapy for Postoperative Cervical Gastric-type Adenocarcinoma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Principal Investigator, Qiu Tang, Chief Physician, Women's Hospital School Of Medicine Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-20250032-R
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Gastric-type Endocervical Adenocarcinoma; Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Paclitaxel; Platinum

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental)
  Interventions: Drug: paclitaxel and platinum
- Control arm (Active Comparator)
  Interventions: Drug: platinum

INTERVENTIONS:
Drug: paclitaxel and platinum — After the start of External Beam Radiation Therapy (EBRT), paclitaxel (150-175 mg/m2) or paclitaxel (albumin-bound) 222-260 mg/m2 + cisplatin (60-75 mg/m2) or carboplatin [Area Under Curve (AUC) = 4-5], Q3W (every 3 weeks is a dosing cycle), administered on the first day of each cycle, for a total of 4 cycles. Adjuvant chemotherapy started 4 weeks after the end of external irradiation therapy, and chemotherapy-related adverse reactions dropped to grade 2 or below before chemotherapy began. If not met, it can be postponed for 2 weeks.
  Arms: Experimental arm
Drug: platinum — During EBRT, cisplatin (40 mg/m2) or carboplatin (AUC = 2) was used for concurrent chemotherapy once a week for a total of 5 times. On the day of cisplatin infusion, radiotherapy should be performed after cisplatin or carboplatin.
  Arms: Control arm

SUMMARY:
Background: Gastric-type endocervical adenocarcinoma (G-EAC) is a new classification of cervical mucinous carcinoma. G-EAC is a unique human papillomavirus unrelated adenocarcinoma that can be distinguished from typical endocervical adenocarcinoma (UEA). In China, adjuvant therapy for cervical cancer after surgery includes not only radiotherapy (RT) or concurrent chemoradiotherapy (CCRT), but also chemotherapy in many cases. However, no previous prospective study has analyzed the adjuvant therapy of G-EAC. This study is the first randomized phase III trial, which aims to recommend better adjuvant treatment options for G-EAC patients at high risk of recurrence in China, in order to better optimize and personalize patient care and improve recurrence-free survival and overall survival.

Methods: This trial is a prospective, multicenter study led by the Department of Radiotherapy, Affiliated Hospital of Obstetrics and Gynecology, Zhejiang University. Recruitment will begin in February 2025, and it is expected that 238 patients with postoperative cervical gastric adenocarcinoma with high risk of recurrence will be recruited from 16 clinical centers in China. Patients will be randomly assigned to the experimental group or the control group in a 1:1 ratio. The experimental group will receive paclitaxel combined with platinum-based concurrent chemoradiotherapy and short-term adjuvant chemotherapy, and the control group will receive the current standard treatment regimen, i.e., platinum-based concurrent chemoradiotherapy, without adjuvant chemotherapy. The primary endpoint of the study is the 2-year progression-free survival, and the secondary endpoints are disease treatment failure pattern, overall survival rate, acute/chronic toxicity incidence, and quality of life assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed Gastric-type endocervical adenocarcinoma;
2. Based on standard examination procedures, it is determined that one of the following risk factors is combined: positive margin, positive paracervical involvement, adnexal involvement, positive lymph nodes, tumor diameter ≥ 4cm, infiltration of the outer 1/3 of the cervical stroma, and vascular tumor thrombus. The specific inclusion can be discussed by two senior clinical doctors;
3. Medical history inquiry and gynecological examination must be performed within 14 days before enrollment to confirm the size of the tumor and International Federation of Gynecology and Obstetrics (FIGO) stage;
4. Chest Computed Tomography (CT) plain scan, abdominal enhanced CT scan, or Positron Emission Tomography (PET)/CT examination within 30 days before enrollment;
5. Pelvic CT, Magnetic Resonance Imaging (MRI) or PET/CT examination within 30 days before enrollment;
6. General condition score 0-1 points;
7. Age 18-65 years old;
8. Laboratory examinations must be performed within 14 days before enrollment, and bone marrow, liver function, and kidney function tests are performed:

   1. White blood cell (WBC) ≥ 3.5 x 10E9/L (normal range)
   2. Neutrophils ≥ 1.5 x 10E9/L;
   3. Platelets ≥ 100 x 10E9/L;
   4. Hemoglobin ≥ 100 g/L (transfusion or other methods are acceptable)
   5. Liver function is within the normal range: alanine aminotransferase (ALT), aspartate aminotransferase (AST) < 1.5 times the upper limit of normal, alkaline phosphatase (ALP) < 2.5 times the upper limit of normal, bilirubin < upper limit of normal.
   6. Renal function is within the normal range: creatinine clearance rate (CCr) > 60 ml/min.

Calculation formula: CCr=(140-age)×weight (kg)/[72×Scr (mg/dl)] or CCr=[(140-age)×weight (kg)]/[0.818×Scr (umol/L)] g) International prothrombin ratio (INR) ≤ 1.5 9. Women of childbearing age must agree to take effective contraceptive measures during the entire treatment study; 10. Patients must sign an informed consent form before enrollment;

Exclusion Criteria:

1. Pathological types of non-gastric adenocarcinomas such as squamous cell carcinoma, adenosquamous carcinoma, undifferentiated carcinoma, small cell carcinoma, neuroendocrine carcinoma, and sarcoma of cervical cancer;
2. Stage IVB;
3. Previous invasive malignant tumors: excluding non-malignant melanoma skin cancer;
4. Systemic chemotherapy in the past 3 years;
5. Previous history of pelvic or abdominal radiotherapy, which may cause overlap of irradiation field for this radiotherapy;
6. Distant metastatic lesions in other organs;
7. The following serious active concurrent diseases:

1) Unstable angina and/or congestive heart failure requiring hospitalization in the past 6 months 2) Transmural myocardial infarction in the past 6 months 3) Acute bacterial or fungal infection requiring intravenous antibiotic treatment at the time of registration 4) Exacerbation of chronic obstructive pulmonary disease or other respiratory diseases requiring hospitalization or hindering the study 5) Jaundice or coagulation disorder caused by poor liver function 6) Acquired immunodeficiency disease (Patients diagnosed with Acquired Immune Deficiency Syndrome (AIDS), or patients suspected of having AIDS who refuse HIV testing); 7) Other immunocompromised states (e.g. organ transplantation, long-term use of glucocorticoids); 8. Pregnant women, breastfeeding women.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
2-year progression-free survival (PFS) | 2 year

SECONDARY OUTCOMES:
Disease failure pattern | 2 year
  The pattern of disease failure will be assessed by the site and number of recurrences or distant metastases.
Overall survival rate | 2 year
Incidence of acute/chronic toxicity | 2 year
Quality of life assessment | 2 year
  Quality of life assessment (time node: 2 years). The patients'quality of life will be assessed using the Quality of Life Questionnaire-Core 30 (QLQ-C30) scale.

IPD SHARING:
Plan to Share IPD: No